CLINICAL TRIAL: NCT00506025
Title: Effectiveness of Cranberry Ingestion on Bacterial Adhesion: Adjunct to Pilot Study of Daily Cranberry Ingestion of Cranberry Juice for the Prevention of Asymptomatic Bacteriuria in Pregnancy
Brief Title: Effectiveness of Cranberry Ingestion on Bacterial Adhesion: An Adjunct Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Deborah A. Wing, Director, Division of Maternal-Fetal Medicine, Obstetrics & Gynecology, University of California, Irvine School of Medicine, University of California, Irvine
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2006-4896
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Results first posted 2010-06-08 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Asymptomatic Bacteriuria
Keywords: Pregnancy; Cranberry; Asymptomatic Bacteruria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cranberry 2xday (Active Comparator): Cranberry juice (C) two times daily, a.m. and p.m.
  Interventions: Dietary Supplement: Cranberry Juice
- Cranberry + Placebo (Active Comparator): De-Activated Cranberry juice in the am, then placebo (P) in the pm
  Interventions: Dietary Supplement: Cranberry Juice
- Placebo 2xday (Placebo Comparator): Placebo in the form of juice two times daily in the a.m. and p.m.
  Interventions: Dietary Supplement: De-Activated Cranberry juice

INTERVENTIONS:
Dietary Supplement: Cranberry Juice — Low-calorie, Low-carbohydrate content 8 oz dose of Cranberry juice
  Arms: Cranberry + Placebo; Cranberry 2xday
Dietary Supplement: De-Activated Cranberry juice — De-Activated Cranberry juice in the am, then placebo (P) in the pm
  Arms: Placebo 2xday

SUMMARY:
This study is to help determine if drinking cranberry juice can decrease risk for asymptomatic bacteriuria (ASB). ASB occurs when there are bacteria in the urine without any symptoms. It will also see if there is a difference in this effect between pregnant and non-pregnant women.This research project is also designed to see what happens to bacterial binding to the lining of the bladder after drinking cranberry juice when special problems occur with pregnancy such as diabetes (a sugar metabolism problem) or ASB is already occurring.

DETAILED DESCRIPTION:
This study is an adjunct to a proposal the premise of which is daily cranberry ingestion during pregnancy may be an effective preventative approach to development of asymptomatic bacteriuria (ASB), a condition which predisposes to both preterm birth and upper urinary tract infection. We proposed to NCCAM a pilot randomized, controlled trial (RCT) in which pregnant women beyond 12 weeks' gestational age will be assigned to one of three schedules for cranberry ingestion: Group A will consume cranberry juice twice a day with breakfast and dinner; Group B will consume cranberry juice at breakfast followed by placebo at dinner; and Group C will consume placebo with meals. Both the cranberry juice and placebo will be of scientific grade, provided by an NIH-contractor. Both are well-characterized, presenting a low-carbohydrate load and low-calorie content per dose (40 cal per 8 oz. dose). Our intent is to 1) generate data comparing the frequency of asymptomatic bacteriuria in pregnant women consuming cranberry juice daily versus placebo, and to 2) create the infrastructure to complete this pilot study and to gather sufficient data to support an R01 for a larger, multi-center RCT focused on the prevention of ASB in pregnancy with daily cranberry juice ingestion.

The reviewers of our proposal enumerated specific weaknesses including 1) a need to evaluate urine from cranberry treated patients, and 2) consideration of bacterial virulence/adherence. The additional variable of gestational diabetes also received comment from the reviewers, and we acknowledge that predisposition in the Hispanic population to this obstetrical complication could impact results. A constituent of cranberries is fructose, which has been implicated in the inhibition of E. coli with type 1 fimbriae (mannose-sensitive) (2). We hypothesize that the glucosuria associated with diabetes in pregnancy may influence the effectiveness of cranberry to prevent asymptomatic bacteriuria.

We must address these weaknesses to strengthen chances for continued funding and competitive renewal.

We have made inquiries with other researchers, and have discovered no direct urine or serum assays by which to measure cranberry metabolites. We understand that there is an R21 proposal under consideration to develop a urinary assay for this purpose under the same RFA. Amy Howell, PhD, of the Marucci Center for Blueberry/Cranberry Research of Rutgers University, one of the field's foremost researchers in this field, and others have indirectly assayed compliance to cranberry by evaluating adherence of piliated E. coli strains before and after cranberry exposure (1). In response to the recent call for proposals for faculty research from the UCI Committee on Research, I proposed this pilot study in collaboration with Dr. Howell.

In this proposal, we will collect the urine from various participants in the R21 trial so as to characterize the effect of cranberry juice ingestion on bacterial adherence. We will ask women to collect their urine for a four-hour time period including first-morning void. The urine samples will be sent to Dr. Howell's laboratory at Rutgers University for analysis. We will collect urine from pregnant women who are assigned to cranberry and to placebo, and from those women who develop bacteriuria following cranberry and following placebo ingestion. We also plan to identify a group of reproductive age, healthy, and non-pregnant women to ingest the active cranberry product or placebo for three days, and on the third day, collect a four-hour timed sample in the same manner as the pregnant women in our control group.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine pregnancy
* Documented fetal viability (either by fetal heart tones present by Doppler auscultation, or by ultrasonic visualization of cardiac motion
* Estimated gestational age by last menstrual period and/or by ultrasonographic fetal measurements of 16 weeks or less

Exclusion Criteria:

* Exclusion criteria will include:
* Suspected non-viable or ectopic gestation
* Patient desires pregnancy termination
* Significant underlying medical complication, such as chronic hypertension, insulin-requiring diabetes, chronic renal failure, cardiac disease, sickle cell disease, etc.
* Maternal age less than 18 years
* Patient is currently on or has received within the two weeks prior to enrollment antimicrobial therapy for reasons other than urinary tract infection.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2006-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Wing, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-seven pregnant women who were enrolled were randomly selected for recruitment into this investigation.
Groups:
- Cranberry 2xday: Cranberry (C) two times daily (C, C; n = 10 pregnant)
- Cranberry + Placebo: Cranberry in the a.m., then placebo (P) in the p.m. (C, P; n = 9 pregnant)
- Placebo 2xday: Placebo two times daily (P, P; n = 8 pregnant)
Period: Overall Study
Arm/Group | Cranberry 2xday | Cranberry + Placebo | Placebo 2xday
Started | 10 | 9 | 8
Completed | 10 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cranberry 2xday | Cranberry + Placebo | Placebo 2xday | Total
Number analyzed (Participants) | 10 | 9 | 8 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 8 | 27
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (5.26) | 27 (5.26) | 24.5 (5.26) | 26.83 (5.263)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 8 | 27
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Activity of Urine From Pregnant Subjects Following Cranberry Juice Cocktail (CJC)
Description: The primary outcome measure was the measurement of bacteriuria in study subject urine, defined as having a urine culture with 100,000 or more of a single uropathogen (measured as cfu per ml).
Time Frame: 7 months, from enrollment at 3 months of pregnancy to delivery
Population: a priori for a pilot study
Measure: Median (Full Range); unit: cfu per ml
Arm/Group | Cranberry 2xday | Cranberry + Placebo | Placebo 2xday
Number analyzed (Participants) | 10 | 9 | 8
cfu per ml | 117.5 [11.0 to 310.0] | 105.0 [41.0 to 385.0] | 110.0 [3.0 to 200.0]

ADVERSE EVENTS:
Arm/Group | Cranberry 2xday | Cranberry + Placebo | Placebo 2xday
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/27

LIMITATIONS AND CAVEATS:
Our study methodology could have been improved with a series of timed urine collections such as collections at pre-treatment, 2, 4 and 6 hours after ingestion of the cranberry juice cocktail and placebo to determine time of maximal effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes